CLINICAL TRIAL: NCT06425185
Title: Differences in Electromyographic Activity of Ankle Stabilizer Muscles in the Different Configurations of a Specific Instability Device: an Observational Study
Brief Title: Differences and Changes in Lower Limb Muscle Activation and Ankle Stability in Different Blackboard Configurations
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rodrigo Martín-San-Agustin, Assistant Professor, University of Valencia
Other Study IDs: 1271077
Record Dates: First submitted 2024-05-12; First posted 2024-05-22 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Electromyography
Keywords: Ankle stability; Muscle activation; Instability device; Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross-sectional study group: The study group consists of 30 subjects who are free from any specific medical condition or injury affecting the lower extremities. These subjects are physically active individuals without any known musculoskeletal disorders or impairments. They all will be assessed in the same way.
  Data collection will take place during single-leg stance on the BB in its different configurations and on the floor. Three attempts of 20 seconds each will be recorded for each condition. The subjects will perform these exercises under the guidance of a trained physiotherapist.
  Interventions: Other: Single-leg stance under different instability conditions

INTERVENTIONS:
Other: Single-leg stance under different instability conditions — Participants will perform three attempts of 20 seconds of single-leg stance on the floor and on the 7 selected configurations of the BB. The order of measurement will be randomized. The description of the chosen configurations can be found in the Detailed Description section. In all cases, the participant's objective is to ensure that the edges of the BB are not in contact with the floor.
  The position of the participant on the BB will be a single-leg stance on the randomly chosen foot, with the contralateral knee slightly flexed and hands placed on the hips. Participants will look at a fixed point placed 3 meters in front of them.
  A rest period of 30 seconds will be allowed between trials. The physiotherapist responsible for supervising the measurements will be the one to adjust the BB configurations when needed.

SUMMARY:
The goal of this observational study is to analyze the differences in muscle activation of six muscles of the lower leg (soleus, gastrocnemius medialis, gastrocnemius lateralis, tibialis anterior, peroneus longus, peroneus brevis) in seven possible configurations of a specific instability device, the Blackboard (BB), as well as on the floor, among healthy active subjects.

The main questions it aims to answer are:

1. Which configuration of the BB produces the highest activation for each studied muscle?
2. Which muscle is the most activated in each configuration of the BB?
3. What is the muscle activation pattern obtained in each configuration of the BB?

A single group of participants will be analyzed. Both the studied leg and the order of configurations of the instability device and ground condition will be randomly assigned. Participants will first undergo a 2-minute continuous walking warm-up, followed by a performance of a maximum voluntary isometric contraction (MVIC) for each muscle, during which the maximum activation produced will be recorded. Each participant will be allowed a 30-second familiarization period on the most unstable configuration of the BB. Three repetitions of 20 seconds will be recorded on both the ground and each configuration, with a 30-second rest between repetitions. The central 10 seconds of each trial will be used for subsequent analysis. The mean of the three repetitions for each muscle will be calculated and subsequently processed and normalized by the maximum activation value during the MIVC.

Finally, a statistical analysis of the differences in muscle activation in each configuration will be conducted with the intention of addressing the mentioned questions.

DETAILED DESCRIPTION:
The use of different instability devices is common in the clinical setting, both for preventive and therapeutic purposes. Numerous studies have demonstrated their effectiveness in improving stability and proprioception, although in most cases in a generalized manner. The need to selectively target specific structures and joints has led to the development of specific instability systems, such as the Blackboard (BB).

The BB is an instability device composed of two rectangular wooden boards, joined together, with Velcro on its base where rounded slats can be freely placed to generate the desired instability according to the patient's or subject's requirements. It is known for its portability, small size, and adaptability, and, as demonstrated in a previous study, similar to traditional devices (BOSU or Wobble board) in activating the Peroneus longus muscle, essential for single-leg stability. However, its detailed functioning is still not fully understood, as the muscle activation it produces during single-leg stance in its different configurations has not been analyzed yet.

This study is a single-group cross-sectional observational study and it will include a sample of 30 participants who will be analyzed in a single session, during single-leg stance on the floor and on the different configurations of the BB. Electrode placement will follow SENIAM guidelines. The session will begin with a 2-minute continuous walking warm-up, followed by the recording of muscle activation in a maximum voluntary isometric contraction (MVIC). Subsequently, the participant will be allowed a 30-second familiarization period on the most unstable configuration of the BB (Total - see description below). Muscle activation of six leg muscles (soleus, medial gastrocnemius, lateral gastrocnemius, tibialis anterior, peroneus longus, and peroneus brevis) will be measured during single-leg stance on the different configurations of the BB and on the ground, randomly.

The analyzed variable will be muscle activation, and the MuscleLab 4020e surface electromyography device from Ergotest Technology AS will be used. The maximum value obtained during the central 10 seconds of the measurement (which will last a total of 20 seconds) will be recorded, in three attempts with 30 seconds of rest between them.

The hypothesis of this study is that by selecting a BB configuration that reinforces the expected muscle function based on ankle biomechanics, its activation will increase. Thus, configurations that require movements such as eversion, to increase activation of the peroneus longus and brevis, or supination, aiming to increase activation of the tibialis anterior, among others, will be analyzed. The description of the different configurations is detailed below, for the right foot:

* Floor: single-leg stance on a firm surface, in this case, the floor
* Rear: single-leg stance on the BB, with the front table fixed and the rear table with the slat placed centrally
* Inver: single-leg stance on the BB, with the front table fixed and the rear table with the slat placed laterally (demanding an inversion movement of the heel)
* Ever: single-leg stance on the BB, with the front table fixed and the rear table with the slat placed medially (demanding an eversion movement of the heel)
* Sup: single-leg stance on the BB, with the rear table fixed and the front table with the slat placed laterally (demanding a supination movement of the forefoot)
* Pro: single-leg stance on the BB, with the rear table fixed and the front table with the slat placed medially (demanding a pronation movement of the forefoot)
* Fore: single-leg stance on the BB, with the rear table fixed and the front table with the slat placed centrally
* Total: single-leg stance on the BB, with both the front and rear tables with the slats placed centrally

In all cases, the subject's objective is to ensure that the edges of the BB are not in contact with the floor.

Thus, the aim of this study is to analyze the differences in electromyographic activity of the six studied muscles across the eight different conditions. This includes identifying the most activated muscles in each condition and determining which condition produces the highest activation of each muscle. Additionally, a secondary aim is to establish patterns of muscular activation for each condition, that is, for each requested movement of the foot and ankle.

ELIGIBILITY:
Inclusion Criteria:

* Not to have experienced lower limb injury or pain within the last year prior to the study
* Self-report as physically active, such that they perform at least 90 minutes of weekly physical activity

Exclusion Criteria:

* Previous participation in any lower limb balance or proprioception exercise program
* The presence of known balance impairments such as vertigo, vestibular or central alterations

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants are being sourced from the Faculty of Physiotherapy of the University of Valencia. They are undergraduate or master's students who have responded to an email invitation sent by one of the professors from the department involved in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
nEMG level of six leg muscles during single-leg stance across eight different conditions | Immediately after the MIVC test, during the single evaluation session, with an approximate duration of 30 minutes (20 minutes of measurement duration, plus time for familiarization and subject preparation)
  The electrode placement area will be shaved and cleaned with alcohol. Muscles analyzed will include soleus, gastrocnemius medialis, gastrocnemius lateralis, tibialis anterior, peroneus longus and peroneus brevis. The MuscleLab 4020e, Ergotest Technology AS surface electromyography device will be used, and adhesive electrode placement will follow SENIAM guidelines.
  Muscle activity will be recorded during 3 periods of 20" with 30" of rest in between. The single-leg stance will be done on the Floor condition and on the 7 instability configurations of the BB.
  The central 10" of the measurement will be used for subsequent analysis. The electromyography signal will be processed and cleaned, and the maximum value registered will be subsequently normalized by the muscle activation obtained during a maximal voluntary isometric contraction, yielding the normalized electromyography (nEMG) for each muscle. The average of the three attempts will be the value used for statistical analysis.

SECONDARY OUTCOMES:
Maximum value of muscle activation of six leg muscles during a maximal voluntary isometric contraction | Immediately after the warm-up, during the single evaluation session, with an approximate duration of 40 minutes (36 minutes of measurement duration, plus time for familiarization and subject preparation)
  The maximum value of muscle activation during a maximal voluntary isometric contraction (MVIC) of the six muscles previously mentioned will be used to normalize the signal collected during the assessment.
  For the peroneus longus, peroneus brevis, and tibialis anterior muscles, this value will be recorded with the participant in supine position, with the examiner resisting eversion and dorsiflexion movements in each case. For the soleus, medial gastrocnemius, and lateral gastrocnemius, the participant will be asked to perform a maximal plantar flexion on one leg, first with the knee slightly flexed and then with the knee extended.
  After a practice trial, each muscle will be tested 3 times, each trial lasting 5", with a 2-minute interval between trials. Verbal encouragement will be provided during testing.
  Finally, the average of the 3 peak values will be used as the maximum reference value for normalization.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Martín-San Agustín, Doctor, Principal Investigator — University of Valencia
Locations (1):
- Rodrigo Martin-San Agustin, Valencia, Spain